CLINICAL TRIAL: NCT00352404
Title: Diagnosis of Intraepithelial Neoplasia in Patients With Long Standing Ulcerative Colitis With Chromoscopic Guided Endomicroscopy
Brief Title: Chromoscopic Guided Endomicroscpy to Diagnose Colitis Associated Dysplasia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DE 000043385
Record Dates: First submitted 2006-07-13; First posted 2006-07-14 (Estimated); Last update posted 2006-07-14 (Estimated); Status verified 2003-08

CONDITIONS: Ulcerative Colitis; Intraepithelial Neoplasia; Cancer
Keywords: Endomicroscopy; Chromoendoscopy; Chromoscopy; Ulcerative Colitis; Intraepithelial Neoplasia
MeSH Terms: conditions — Colitis, Ulcerative; Carcinoma in Situ; Neoplasms

INTERVENTIONS:
Device: Endomicroscope

SUMMARY:
Timely diagnosis of intraepithelial neoplasias (premalignant condition)is of crucial importance for clinical management of ulcerative colitis. We assessed the value of combined chromoscopy and endomicroscopy for diagnosis of intraepithelial neoplasias in a randomised controlled trial.

Endomicroscopy is a new device which enables microscopy of the mucosal layer during ongoing colonoscopy. Chromoscopy means topical staining of mucosal surface to unmask areas of interest, which are subsequently examined with the endomicroscopic system.

DETAILED DESCRIPTION:
Ulcerative colitis (UC) is an immune cell-mediated inflammatory bowel disease characterized by mucosal ulcerations, rectal bleeding, diarrhea, and abdominal pain. Patients with long standing UC face an increased risk for development of colitis associated colorectal cancer. Factors associated with increased risk for cancer development include the duration of the disease, extensive colonic involvement (pancolitis, backwash ileitis), primary sclerosing cholangitis and severe chronic active inflammation. Based on these observations, colonoscopic surveillance in patients with long-standing UC is highly recommended.

The main objective of surveillance colonoscopy in UC is to detect neoplasia at a surgically curative and preferably pre-invasive stage. However, in contrast to sporadic colorectal cancer, the growing pattern of neoplastic tissue in UC is often flat and multifocal. Therefore, significant lesions during conventional colonoscopy in UC are frequently overlooked. Chromoscopy with topically applied dyes such as methylene blue or indigo carmine facilitates the endoscopic detection of flat, circumscribed colitis associated neoplastic changes in UC. In fact, five controlled studies showed that the diagnostic yield for the detection of intraepithelial neoplasia (IN) using chromoscopy is higher as compared to conventional colonoscopy with random biopsies. Based on the above studies, chromoscopy has recently been considered for incorporation into US guidelines for surveillance of patients with long-standing UC. However, although this technique does allow identification of mucosal lesions, it is not suitable for accurate endoscopic diagnosis of intraepithelial neoplasias in UC due to the lack of cellular resolution and subsurface imaging. For endoscopy, novel techniques allowing accurate diagnoses during ongoing examination are highly desirable and may allow appropriate and immediate therapeutic manoeuvres (e.g. resection versus biopsy). Recently, a miniaturized confocal microscope has been developed integrated in the distal tip of a conventional colonoscope . This new diagnostic technology for gastrointestinal endoscopy, denoted confocal endomicroscopy, enables histological evaluation of the mucosal layer during ongoing colonoscopy. Furthermore, in patients screened for sporadic colorectal cancer, surface and subsurface analysis at cellular and subcellular resolution can be used to predict intraepithelial neoplasias (INs) with high accuracy. However, due to the time required for examination of large surface areas, this technique is not suitable for screening of the entire colonic surface in UC to detect neoplasias in flat mucosa.

In the present study, we employ chromoscopy to identify potential neoplastic lesions and combine this for the first time with endomicroscopy for the endoscopic diagnosis of colitis associated intraepithelial neoplasias in UC. Using such chromoscopy guided endomicroscopy we will ecaluate whether the diagnostic yield diagnosing IN can be significantly increased.

ELIGIBILITY:
Inclusion Criteria:

* Clinically and histologically verified UC
* Disease duration >8 years
* Colitis Activity Index ≤8
* Activity index of Truelove and Witts: mild

Exclusion Criteria:

* Known intraepithelial neoplasia or colorectal cancer
* Coagulopathy (Prothrombin time <50% of control, Partial thromboplastin time >50 s)
* Impaired renal function (Creatinine >1.2 mg/dL)
* Pregnancy or breast feeding
* Inability to obtain informed consent
* Known allergy to methylene blue or Fluorescein

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114
Dates: Start 2003-08; Study Completion 2004-11

PRIMARY OUTCOMES:
Histological proof of neoplastic tissue (Intraepithelial neoplasia or cancer)

SECONDARY OUTCOMES:
Prediction of extent and severity of inflamed mucosa

CONTACTS AND LOCATIONS:
Overall Officials: Peter R. Galle, MD PhD, Study Director — Johannes Gutenberg University, Germany
Locations (1):
- I. Med. Klinik, Johannes Gutenberg Universitaet, Mainz, Rhineland-Palatinate, Germany

REFERENCES:
- See also: Information about the new device — http://www.endomicroscopy.com